CLINICAL TRIAL: NCT03145233
Title: Isometric Versus Isotonic Exercise for Greater Trochanteric Pain Syndrome - a Randomised Controlled Trial Comparing Two Rehabilitation Programmes
Brief Title: Isometric Versus Isotonic Exercise for Greater Trochanteric Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN17PY175
Record Dates: First submitted 2017-04-25; First posted 2017-05-09 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Gluteal Tendinitis
Keywords: physiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric exercise (Experimental): 12 week Isometric exercise programme - two exercises (one side-lying and the other standing); six repetitions of each with muscle contraction sustained for 30 seconds. Exercises performed once daily with each session lasting no longer than 10 minutes.
  Interventions: Other: Isometric exercise programme
- Isotonic exercise (Experimental): 12 week Isotonic exercise programme - two exercises (one side-lying and the other standing); each exercise - 3 sets of 10 repetitions, each repetition 6 seconds duration. Exercises performed once daily with each session lasting no longer than 10 minutes.
  Interventions: Other: Isotonic exercise programme

INTERVENTIONS:
Other: Isometric exercise programme — Exercise programme where the muscle length and joint angle do not change due to the limb being held in a static position
  Arms: Isometric exercise
Other: Isotonic exercise programme — Exercise programme where both the muscle length and joint angle do change, consisting of concentric muscle actions (where the muscle shortens) and eccentric muscle actions (where the muscle lengthens)
  Arms: Isotonic exercise

SUMMARY:
This pilot randomised controlled trial will directly compare the effect of isometric exercise to isotonic exercise over a period of 12 weeks for participants with a clinical diagnosis of Greater Trochanteric Pain Syndrome (GTPS).

DETAILED DESCRIPTION:
Pain at the side of the hip over or around the greater trochanter of the femur has previously been termed as Greater Trochanteric Pain Syndrome (GTPS). Recent research has found that it is normally due to the gluteal tendons being torn or injured and is often termed as 'gluteal tendinopathy'. GTPS predominantly affects adults aged 40-60 years and is the second most common condition affecting the hip region after osteoarthritis. Quality of life scores are similar to those with advanced hip osteoarthritis but despite its prevalence and disease burden the most effective treatment for this problem is currently unknown.

Numerous studies have shown that exercise programmes are the most effective treatment for other lower limb tendon problems, particularly the Achilles and patella. These programmes typically last a minimum of 12 weeks and are often prescribed by physiotherapists as first-line treatment. However, there is currently limited evidence to support exercise for gluteal tendinopathy. The study plans to directly compare two different types of exercise programmes for those with GTPS for a period of 12 weeks. One group will receive an isometric exercise programme (where the muscle length does not change) and a second group an isotonic exercise programme (where the muscle length does change).

The primary outcome measure which will be used has recently been validated for patients with gluteal tendinopathy and measures function and disability. Additional secondary outcome measures will evaluate aspects relating to quality of life, physical activity and pain. Both groups will be compared at the start of the study and at different times up to a maximum of 12 weeks to help determine if one exercise programme is better than the other.

The results of this pilot study will also help to identify whether a larger trial would be possible in the future.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent
* Lateral hip pain for greater than 3 months
* Pain on direct palpation of the gluteal tendon insertion on the greater trochanter and additionally at least one of the following pain provocation tests must also be positive:

  1. FABER (Flexion, Abduction, External Rotation of the hip)
  2. FADER (Flexion, Adduction, External Rotation of the hip)
  3. FADER and resisted Internal Rotation (IR) (FADER position plus resisted IR of the hip)
  4. Single leg stand for 30 seconds
  5. Resisted hip abduction at end-range adduction

Exclusion Criteria:

* Physiotherapy for lateral hip pain in the past 6 months
* Corticosteroid injection for lateral hip pain in past 3 months
* Inability to actively abduct hip in side-lying
* Pain reproduced with FADIR (Flexion, Adduction, Internal Rotation of hip) with concurrent hip osteoarthritis on anteroposterior (AP) pelvis x-ray defined as Kellgren-Lawrence > Grade 2 (mild)
* Previous hip or lumbar spine surgery in past 12 months
* Inflammatory joint disease
* Unstable diabetes or cardiovascular disease
* Known neurological disorders
* Widespread chronic pain or fibromyalgia
* Avascular necrosis
* Pregnancy
* Participants unable or unwilling to give informed consent
* Participants who are unable to write, read or comprehend English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Measure of disability | Baseline, 4 weeks and 12 weeks
  Change in score on Victorian Institute of Sport Assessment-Gluteal (VISA-G) questionnaire

SECONDARY OUTCOMES:
Quality of Life | Baseline, 4 weeks and 12 weeks
  Change in score on European Quality of Life (EQ-5D-5L) questionnaire
Perceived change in hip pain | Baseline, 4 weeks and 12 weeks
  Change in score on Global Rating of Change (GROC) Scale
Pain intensity | Baseline, 4 weeks and 12 weeks
  Change in score on Numeric Pain Rating Scale (NPRS)
Pain catastrophisation | Baseline, 4 weeks and 12 weeks
  Change in score on Pain Catastrophising Scale
Hip disability | Baseline, 4 weeks and 12 weeks
  Change in score on Hip Disability and Osteoarthritis Outcome Score (HOOS)
Physical activity | Baseline, 4 weeks and 12 weeks
  Change in score on International Physical Activity Questionnaire Short Form (IPAQ-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Millar, PhD FRCSEd, Study Director — University of Glasgow; Lorna Paul, MPhil PhD, Study Director — Glasgow Caledonian University
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No